CLINICAL TRIAL: NCT00054327
Title: Hematopoietic Stem Cell Transplantation Using Bone Marrow Or Peripheral Blood Stem Cells From Matched, Unrelated, Volunteer Donors
Brief Title: Donor Stem Cell Transplant in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1Y00; P30CA043703 (NIH); CASE-CWRU-1Y00 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Results first posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: adult acute myeloid leukemia in remission; childhood acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 3 follicular lymphoma; secondary acute myeloid leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent mantle cell lymphoma; refractory anemia with ringed sideroblasts; refractory anemia; chronic myelomonocytic leukemia; refractory cytopenia with multilineage dysplasia; previously treated myelodysplastic syndromes; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes; relapsing chronic myelogenous leukemia; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; juvenile myelomonocytic leukemia; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Anemia, Refractory; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Leukemia, Myelomonocytic, Juvenile; Congenital Abnormalities | interventions — Busulfan; Cyclophosphamide; Cytarabine; Radiotherapy; Whole-Body Irradiation; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Regimen A (Experimental): Patients receive cytarabine 3.0gm/M² IV over 1 hour twice daily on days -9 to -7 and cyclophosphamide 45mg/kg IV over 2 hours on days -6 and -5. Patients also undergo total body irradiation (TBI), 165 cGY, twice daily on days -4 to -1 for a total of 1320 cGY.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Radiation: radiation therapy; Procedure: Stem Cell Transfusion
- Regimen B-1 (Experimental): Patients receive cyclophosphamide 60 mg/kg IV on days -6 and -5. Patients also undergo total body irradiation (TBI) twice daily on days -4 to -1 for a total of 1320 cGY..
  Interventions: Drug: cyclophosphamide; Radiation: radiation therapy; Procedure: Stem Cell Transfusion
- Regimen B-2 (Experimental): Patients receive cyclophosphamide 60 mg/kg IV over 2 hours on days -5 and -4. Patients also undergo TBI twice daily on days -3 to -1 for a total of 1200 cGY.
  Interventions: Drug: cyclophosphamide; Radiation: radiation therapy; Procedure: Stem Cell Transfusion
- Regimen C (Experimental): Patients receive oral busulfan 1mg/kg/dose (or 40mg/m2/dose for young children)4 times daily on days -8 to -5 and cyclophosphamide 60 mg/kg IV over 2 hours on days -4 to -2.
  Interventions: Drug: busulfan; Drug: cyclophosphamide; Procedure: Stem Cell Transfusion
- Regimen B-3 (Experimental): Patients undergo total body irradiation (TBI) twice daily on days -7 to -5 for a total of 1200 cGY. Patients then receive cyclophosphamide 60 mg/kg IV on days -4 and -3.
  Interventions: Drug: cyclophosphamide; Radiation: radiation therapy; Procedure: Stem Cell Transfusion
- Regimen D (Experimental): Patients receive total body irradiation (TBI) on days T -6, -5 and -4 for a total of 1320 cGy , then etoposide (60mg/kg/dose) on day -3.
  Interventions: Radiation: radiation therapy; Drug: Etoposide; Procedure: Stem Cell Transfusion

INTERVENTIONS:
Drug: busulfan — Given orally 1mg/kg/dose (or 40mg/m2/dose for young children)
  Other Names: Myleran
  Arms: Regimen C
Drug: cyclophosphamide — Given IV
  Other Names: cytoxan; CTX; CPM
  Arms: Regimen A; Regimen B-1; Regimen B-2; Regimen B-3; Regimen C
Drug: cytarabine — Given IV
  Other Names: Cytosine Arabinoside; Cytosar-U; Ara-C; Arabinosyl
  Arms: Regimen A
Radiation: radiation therapy — Patients undergo total body irradiation
  Other Names: Total body irradiation
  Arms: Regimen A; Regimen B-1; Regimen B-2; Regimen B-3; Regimen D
Drug: Etoposide — infusion
  Other Names: VP-16; VePesid®; VP-16-213; EPEG; epipodophyllotoixn
  Arms: Regimen D
Procedure: Stem Cell Transfusion

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor peripheral stem cell transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the stem cells from a related donor, that do not exactly match the patient's blood, are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

PURPOSE: This phase II trial is studying how well giving chemotherapy with or without radiation therapy followed by donor stem cell transplant works in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine a standard approach to hematopoietic stem cell transplantation with matched unrelated donors in patients with hematologic malignancies.
* Determine the toxicity of this regimen in these patients.
* Determine the relapse rate and survival rate in patients treated with this regimen.
* Correlate incidence and severity of graft-versus-host disease with relapse and survival in patients treated with this regimen.

OUTLINE: Patients receive 1 of the following preparative regimens:

* Regimen A: Patients receive cytarabine IV over 1 hour twice daily on days -9 to -7 and cyclophosphamide IV over 2 hours on days -6 and -5. Patients also undergo total body irradiation (TBI) twice daily on days -4 to -1.
* Regimen B-1: Patients receive cyclophosphamide IV and TBI as in regimen A.
* Regimen B-2: Patients receive cyclophosphamide IV over 2 hours on days -5 and -4. Patients also undergo TBI twice daily on days -3 to -1.
* Regimen B-3: Patients receive TBI on days -7 to -5. Patients receive cyclophosphamide IV over on days -4 to -3.
* Regimen C: Patients receive oral busulfan 4 times daily on days -8 to -5 and cyclophosphamide IV over 2 hours on days -4 to -2.
* Regimen D: Patients receive TBI on days -6 to -4. Patients receive etoposide infusion on day -3.

All patients undergo stem cell transplantation from a matched, unrelated donor on day 0.

Patients are followed weekly for 100 days, at 6 months, and then every 6 months for 2.5 years.

PROJECTED ACCRUAL: 50

ELIGIBILITY:
Eligibility Criteria:

1. Patients with histologic confirmation of the following diseases are eligible:

   1. AML in first, second or greater remission
   2. AML in early relapse, defined at <30% marrow blasts
   3. ALL in second or greater complete remission
   4. High risk ALL in first complete remission, with high risk being defined by the presence of t(4;11), t(9;22), or t(8;14) translocation, or patients presenting with extreme hyperleukocytosis (initial WBC >500 K/ml) or failure to achieve a complete remission after standard induction therapy.
   5. CML
   6. Myelodysplastic syndromes (including evolution to AML, e.g., Refractory Anemia with Excess Blasts (RAEB), or Refractory Anemia with Excess Blasts in transformation (RAEB-t).
   7. Lymphoma (intermediate and high grade) chemosensitive (CR or PR) after first or greater relapse or chemosensitive to first line therapy but only achieving PR.
   8. Hematologic Disease and Inherited Immunodeficiencies
   9. Hodgkin's disease, relapsed or refractory to standard treatments.
2. Patients must be less than or equal to 55 years of age.
3. Patients (or guardians if minor) must be able to give informed consent. Children older than 11 years of age must assent to the process.
4. Patients or their guardians must demonstrate proof-of-payment.
5. Patients must have an ECOG Performance Status of 2 or less. (See Appendix I)
6. Patients must have no evidence of active infection at the time of transplantation.
7. Patients must be HIV nonreactive.
8. Patients must have a pre-transplant, multi-organ assessment prior to transplantation with the following outcome:

   1. resting ejection fraction of 50% or greater (or shortening fraction greater than 28% for small children).
   2. Diffusion capacity of 50% or greater of predicted, a FEV1 of 50% or greater, and a P2O of 80 mm Hg as demonstrated on pulmonary function testing.
   3. serum creatinine of less than or equal to 2.0 mg/dL and/or a corrected creatinine clearance of 50 ml/min or greater on 24 hr urine.
   4. A total bilirubin of less than 2.5 mg/dL and an AST less than 4 times the upper limits of normal.
9. Females who are childbearing age may not be pregnant or lactating and must have a current negative pregnancy test

Ineligibility Criteria:

* Patients who have a life expectancy of less than three months with therapy.
* Patients who have an ECOG performance status greater than 2, (See Appendix I) or Lansky Scale < 70%.
* Patients who have angina and/or congestive heart failure requiring treatment, or who have had a myocardial infarction within the past year.
* Patients who have a resting ejection of less than 50% (or shortening fraction less than 28%) and who have not been cleared for transplant by cardiology
* Patients who have severe renal disease as demonstrated by a serum creatinine greater than 2.0 mg/dL and/or a corrected creatinine clearance less than 50 ml/min. (corrected for BSA of 1.73 m¬2)
* Patients who have had any complication that makes the risk of death during transplantation from non-malignant causes greater than the risk of relapse.
* Patients who have any active infection such as a soft tissue infection, sinus infection, dental infection, fungal infection or hepatitis including chronic active hepatitis; if the infection is successfully treated, the patient may be reconsidered for transplantation at a later date.
* Patients who have decreased pulmonary function due to any disorder as demonstrated by a diffusion capacity of less than 50% of predicted, a FEV1 of less than 50% of predicted or a PO2 of less than 80 mm Hg pulmonary function testing.
* Patients who have decreased liver function as demonstrated by a total bilirubin of greater than 2.5 mg/dL and/or an AST greater than 4 times the upper limits of normal.
* Patients who have diabetes mellitus will be considered on a case-by-case basis. However, patients with diabetes who are not controlled by medical management will be ineligible.

-Patients who have a significant psychiatric illness will be considered on a case- by-case basis. With the patient's consent, their Mental Health Care worker will assist the managing transplant physicians in determining if the patient can safely undergo transplantation and comply with followup recommendations.

* Psychosocial assessment by the bone marrow transplant team may identify individuals for whom this form of therapy may be contraindicated. This decision will be based upon estimated adequacy of patient support systems and prediction of patient's compliance with medications, required diagnostic procedures and/or follow-up care.
* Females who are childbearing age may not be pregnant or lactating and must have a current negative pregnancy test
* Patients who had a stem cell transplant less than one year earlier

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2000-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cooke, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-five patients were recruited from local medical clinic from November 2000 through November 2009.One patient relapsed and never received a transplant.
Period: Overall Study
Arm/Group | Regimen A | Regimen B-1 | Regimen B-2 | Regimen B-3 | Regimen C | Regimen D
Started | 11 | 4 | 3 | 4 | 10 | 2
Completed | 10 | 4 | 3 | 4 | 10 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Engraftment failure | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A | Regimen B-1 | Regimen B-2 | Regimen B-3 | Regimen C | Regimen D | Total
Number analyzed (Participants) | 11 | 4 | 3 | 4 | 10 | 2 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 4 | 0 | 1 | 0 | 0 | 13
  Between 18 and 65 years | 3 | 0 | 3 | 3 | 10 | 2 | 21
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 3 | 5 | 1 | 16
  Male | 7 | 2 | 2 | 1 | 5 | 1 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 11 | 3 | 3 | 4 | 10 | 2 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 11 | 4 | 3 | 4 | 10 | 2 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rates of Durable Engraftment
Description: Number of days that patients take to reach engraftment defined as time to hematologic engraftment will be defined as ANC >500/µl and platelets >20K/µl without transfusion support.
Time Frame: at day 42
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Regimen A | Regimen B-1 | Regimen B-2 | Regimen B-3 | Regimen C | Regimen D
Number analyzed (Participants) | 10 | 4 | 3 | 4 | 10 | 2
days | 17.9 (5.801341) | 15.75 (6.946222) | 13 (3) | 18.25 (4.573474) | 13.9 (5.237684) | 10.5 (0.707107)

2. Secondary Outcome: Graft-versus-host Disease (GVHD)
Description: Number of patients that develop acute graft-versus-host disease by grades 0-4. Grade O is no development of GVHD. Grade 1-4 is increase severity of skin, liver and gut involvement with 1 being least severe and 4 being most severe.
Time Frame: at 100 days post transplant
Measure: Number; unit: participants
Arm/Group | Regimen A | Regimen B-1 | Regimen B-2 | Regimen B-3 | Regimen C | Regimen D
Number analyzed (Participants) | 10 | 4 | 3 | 4 | 10 | 2
participants
  Grade 0 | 0 | 1 | 1 | 1 | 1 | 0
  Grade 1 | 2 | 1 | 0 | 0 | 1 | 0
  Grade 2 | 6 | 2 | 1 | 0 | 5 | 0
  Grade 3 | 2 | 0 | 0 | 3 | 3 | 0
  Grade 4 | 0 | 0 | 1 | 0 | 0 | 2

3. Secondary Outcome: Incidence of Recurrent Disease
Description: Number of patients that have disease recurrence.
Time Frame: at day 100 post transplant
Measure: Number; unit: participants
Arm/Group | Regimen A | Regimen B-1 | Regimen B-2 | Regimen B-3 | Regimen C | Regimen D
Number analyzed (Participants) | 10 | 4 | 3 | 4 | 10 | 2
participants | 4 | 2 | 0 | 1 | 2 | 0

4. Secondary Outcome: Toxicity as Measured by CTC v2.0
Description: Number of patients that experience grade 3 or above toxicity. See serious adverse event list for toxicities.
Time Frame: at 100 days post transplant
Measure: Number; unit: participants
Arm/Group | Regimen A | Regimen B-1 | Regimen B-2 | Regimen B-3 | Regimen C | Regimen D
Number analyzed (Participants) | 11 | 4 | 3 | 4 | 10 | 2
participants | 0 | 0 | 1 | 2 | 2 | 0

5. Post Hoc Outcome: Number of Patients With Overall Survival at 2 Years.
Time Frame: at 2 years from transplant
Measure: Number; unit: participants
Arm/Group | Regimen A | Regimen B-1 | Regimen B-2 | Regimen B-3 | Regimen C | Regimen D
Number analyzed (Participants) | 11 | 4 | 3 | 4 | 10 | 2
participants | 5 | 2 | 2 | 1 | 5 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected while patients were on study over a an eleven year period. Only grade 3 and above toxicity were collected.
Description: "0" Total Number of Participants at Risk (e.g.., other [non-serious] adverse events were not collected or assessed as part of the study).
Arm/Group | Regimen A | Regimen B-1 | Regimen B-2 | Regimen B-3 | Regimen C | Regimen D
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/4 | 1/3 | 2/4 | 2/10 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A (N=11) | Regimen B-1 (N=4) | Regimen B-2 (N=3) | Regimen B-3 (N=4) | Regimen C (N=10) | Regimen D (N=2)
Melena/GI bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Elevated Bilirubin associated with graft versus host disease (GVHD) (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Memory loss (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Edema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mood alteration-anxiety, agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Death not associated with CTCAE term - Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes